CLINICAL TRIAL: NCT05016544
Title: A Phase Ib Clinical Study Evaluating the Safety and Efficacy of Inetetamab in Combination With Pyrotinib in HER2 Mutant or Amplified Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Inetetamab in Combination With Pyrotinib in HER2 Mutant or Amplified Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-191
Record Dates: First submitted 2021-08-08; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Inetetamab; Pyrotinib; HER2-activated mutation; HER2-amplification
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Sequential assignment by traditional 3+3 dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inetetamab+Pyrotinib (Experimental): Dose Escalation and Dose Expansion: Inetetamab in combination with Pyrotinib in HER2 mutant or amplified participants with advanced or metastatic NSCLC
  Interventions: Drug: inetetamab; Drug: Pytotinib

INTERVENTIONS:
Drug: inetetamab — All dose levels will receive 8 mg/kg loading dose for cycle 1, followed by 6 mg/kg in subsequent cycles, every 3 weeks.
Drug: Pytotinib — Starting pytotinib Dose of 240mg:
  Cohort 1: pyrotinib 240mg p.o. d1 to d21, q3w; Cohort 2: pyrotinib 320mg p.o. d1 to d21, q3w; Cohort 3: pyrotinib 400mg p.o. d1 to d21, q3w.

SUMMARY:
This is a Phase 1, open-label study to evaluate the safety and the efficacy of inetetamab in combination with pyrotinib in patients in HER2 mutant or amplified patients with advanced non-small cell lung cancer

DETAILED DESCRIPTION:
This study is a multi-center, opening, dose-escalating phase Ib clinical trial. The aim of the study is to evaluate the safety and efficacy of inetetamab combined with pyrotinib in the treatment of patients in HER2 mutant or amplified patients with advanced non-small cell lung cancer .Primary endpoint of the study is dose-limiting toxicity dosage and safety. Efficacy indicators including objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), overall survival (OS) are as Secondary endpoint. Up to 48 NSCLC patients will be enrolled the treatment will be performed 3+3 dose-escalation phase I design and expanded to phase II study. A treatment cycle lasts 3 weeks,and the combined medication will be continued until the occurrence of toxicity intolerance,disease progression,or death,or patients refuse to continue participating in this clinical study,or the investigators determine that the medication must be terminated.

The recommended initial consistent dose of inetetamab in groups 1-3 are 8 mg/kg, intravenous infusion for more than 90 minutes, and the maintenance dose is 6 mg/kg.

The oral doses of pyrotinib in groups 1-3 were 240 mg, 320 mg, or 400 mg, respectively.

Safety evaluation will be taken according to hematological toxicity, non-hematological toxicity and National Cancer Institute (NCI)-Common Terminology Criteria (CTC) For Adverse Events (AE) V5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18;
2. Histologically or cytologically documented metastatic NSCLC, HER2 activation amplification or mutation stage IIIB-IV NSCLC patient;
3. At least 1 measurable lesion according to RECIST 1.1;
4. ECOG score 0 or 1;
5. Life expectancy of at least 3 months;
6. Within one week before admission, blood routine examination was basically normal:

   1. hemoglobin ≥90g/L or ≥5.6mmol/L;
   2. neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L;
   3. platelet count (PLT) ≥ 100 × 10 ^ 9 / L;
   4. Liver and kidney function tests were basically normal within one week before enrollment;
   5. total bilirubin (TBIL) ≤ 1.5 × upper limit of normal value (ULN);
   6. alanine aminotransferase (ALT / AST) ≤ 2.5 × ULN (liver metastasis patients ≤ 5xuln);
   7. serum creatinine ≤ 1.5 × ULN;
   8. Partially activated thrombin time(APTT)≤ 1.5 × ULN;
7. For fertile women had negative blood pregnancy tests 7 days before screening;
8. willing to participate and sign the informed consent in person.

Exclusion Criteria:

1. Patients who have received anti-HER2 monoclonal antibody therapy;
2. Have received chemotherapy, biotherapy, targeted therapy, immunotherapy and other anti-tumor therapies within 4 weeks prior to the first use of the study drug including: oral small molecule targeted drugs within 2 weeks prior to the first use of the study drug or within 5 half-lives of known drugs (depending on the time);Radiotherapy was performed within 2 weeks prior to the first administration of the study drug;
3. Have received other clinical study drugs within 4 weeks prior to the first study drug administration;
4. Patients who underwent major surgery within 4 weeks prior to the first dosing of the study drug(except needle biopsy or significant trauma);
5. Those who have been known to have allergic history to the drug components of this regimen;
6. Study drugs that had used a CYP3A4 inhibitor, inducer, or a narrow therapeutic window with a CYP3A4-sensitive substrate ,P-ep strong inducer and inhibitor within 14 days before first administration;
7. The adverse reactions of previous antitumor therapy have not recovered to CTCAE 5.0 grade 1(Hair loss and other toxicities were excluded for which the researchers judged no safety risk);
8. Patients with central nervous system metastasis and clinical symptoms;
9. History of immunodeficiency, including positive HIV test, or suffering from other acquired, congenital immunodeficiency diseases, or history of organ transplantation;
10. Active hepatitis B (HBV virus titer 1000 copies /ml or 200IU/ml);Hepatitis C virus, syphilis infection;
11. Severe heart disease or discomfort, including, but not limited to, the following: complete left bundle branch block or degree atrioventricular block, history of myocardial infarction, angioplasty, coronary artery bridging, patients with prolonged QT/QTc interval at baseline (QTcF men >450 ms, women >480ms), significant ventricular arrhythmias (such as ventricular tachycardia), history of heart failure or systolic dysfunction (LVEF < 50%), cardiac failure, New York College of Cardiology (NYHA) grade II or higher, uncontrolled hypertension (systolic blood pressure > 180 mmHg ), history or current history of cardiomyopathy that the investigator judged to have an impact on the study;
12. Inability to swallow medications orally, or that the investigator determines severely affect gastrointestinal absorption;
13. Other malignant tumors in the past 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma or in situ cervical cancer and/or breast cancer;
14. Any history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring steroid treatment, or evidence of clinically active interstitial lung disease;
15. Patients with a history of other serious systemic diseases who were judged by the investigator to be unsuitable for clinical trials;
16. Alcohol or drug dependence;
17. Have a clear history of neurological or mental disorders, including epilepsy or dementia;
18. Pregnant and/or breastfeeding;
19. Any other reason the investigator considers the patient is not suitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Dose escalation | Up to 21 days after the first dose
  Number of Participants with a Dose-Limiting Toxicity (DLT)
Incidence of adverse events | Up to 30 days after the last dose of inetetamab or pyrotinib
  Incidence, severity, and serious adverse events (SAEs) based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

SECONDARY OUTCOMES:
Objective response rate | up to12 months
  Per RECIST v1.1 criteria, the proportion of patients whose best remission was CR or PR accounted for the total number of evaluable patients.
Disease Control Rate | up to12 months
  Per RECIST v1.1 criteria, the proportion of patients whose best remission was CR , PR and SD accounted for the total number of evaluable patients.
Progression free survival | 24 months
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Overall survival | 36 months
  Overall survival (OS) is defined as the time from the date of first dosing till death due to any cause.
Investigation on molecular markers associated with the clinical efficacy and the mechanism of drug resistance | 36 months
  Using next generation sequencing (NGS) method to detect 22 genes from circulating free DNA (cf-DNA) in patients, periphereal blood sample were collected at baseline, first time tumor efficacy evaluation, and withdrawn study due to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cocco E, Lopez S, Santin AD, Scaltriti M. Prevalence and role of HER2 mutations in cancer. Pharmacol Ther. 2019 Jul;199:188-196. doi: 10.1016/j.pharmthera.2019.03.010. Epub 2019 Apr 2. PMID 30951733
- [Result] Pisters KM, Le Chevalier T. Adjuvant chemotherapy in completely resected non-small-cell lung cancer. J Clin Oncol. 2005 May 10;23(14):3270-8. doi: 10.1200/JCO.2005.11.478. PMID 15886314
- [Result] Bonomi PD. Implications of key trials in advanced nonsmall cell lung cancer. Cancer. 2010 Mar 1;116(5):1155-64. doi: 10.1002/cncr.24815. PMID 20087963
- [Result] Stephens P, Hunter C, Bignell G, Edkins S, Davies H, Teague J, Stevens C, O'Meara S, Smith R, Parker A, Barthorpe A, Blow M, Brackenbury L, Butler A, Clarke O, Cole J, Dicks E, Dike A, Drozd A, Edwards K, Forbes S, Foster R, Gray K, Greenman C, Halliday K, Hills K, Kosmidou V, Lugg R, Menzies A, Perry J, Petty R, Raine K, Ratford L, Shepherd R, Small A, Stephens Y, Tofts C, Varian J, West S, Widaa S, Yates A, Brasseur F, Cooper CS, Flanagan AM, Knowles M, Leung SY, Louis DN, Looijenga LH, Malkowicz B, Pierotti MA, Teh B, Chenevix-Trench G, Weber BL, Yuen ST, Harris G, Goldstraw P, Nicholson AG, Futreal PA, Wooster R, Stratton MR. Lung cancer: intragenic ERBB2 kinase mutations in tumours. Nature. 2004 Sep 30;431(7008):525-6. doi: 10.1038/431525b. PMID 15457249
- [Result] Arcila ME, Chaft JE, Nafa K, Roy-Chowdhuri S, Lau C, Zaidinski M, Paik PK, Zakowski MF, Kris MG, Ladanyi M. Prevalence, clinicopathologic associations, and molecular spectrum of ERBB2 (HER2) tyrosine kinase mutations in lung adenocarcinomas. Clin Cancer Res. 2012 Sep 15;18(18):4910-8. doi: 10.1158/1078-0432.CCR-12-0912. Epub 2012 Jul 3. PMID 22761469
- [Result] Gatzemeier U, Groth G, Butts C, Van Zandwijk N, Shepherd F, Ardizzoni A, Barton C, Ghahramani P, Hirsh V. Randomized phase II trial of gemcitabine-cisplatin with or without trastuzumab in HER2-positive non-small-cell lung cancer. Ann Oncol. 2004 Jan;15(1):19-27. doi: 10.1093/annonc/mdh031. PMID 14679114
- [Result] Lara PN Jr, Laptalo L, Longmate J, Lau DH, Gandour-Edwards R, Gumerlock PH, Doroshow JH, Gandara DR; California Cancer Consortium. Trastuzumab plus docetaxel in HER2/neu-positive non-small-cell lung cancer: a California Cancer Consortium screening and phase II trial. Clin Lung Cancer. 2004 Jan;5(4):231-6. doi: 10.3816/clc.2004.n.004. PMID 14967075
- [Result] Perera SA, Li D, Shimamura T, Raso MG, Ji H, Chen L, Borgman CL, Zaghlul S, Brandstetter KA, Kubo S, Takahashi M, Chirieac LR, Padera RF, Bronson RT, Shapiro GI, Greulich H, Meyerson M, Guertler U, Chesa PG, Solca F, Wistuba II, Wong KK. HER2YVMA drives rapid development of adenosquamous lung tumors in mice that are sensitive to BIBW2992 and rapamycin combination therapy. Proc Natl Acad Sci U S A. 2009 Jan 13;106(2):474-9. doi: 10.1073/pnas.0808930106. Epub 2009 Jan 2. PMID 19122144
- [Result] Shimamura T, Ji H, Minami Y, Thomas RK, Lowell AM, Shah K, Greulich H, Glatt KA, Meyerson M, Shapiro GI, Wong KK. Non-small-cell lung cancer and Ba/F3 transformed cells harboring the ERBB2 G776insV_G/C mutation are sensitive to the dual-specific epidermal growth factor receptor and ERBB2 inhibitor HKI-272. Cancer Res. 2006 Jul 1;66(13):6487-91. doi: 10.1158/0008-5472.CAN-06-0971. PMID 16818618
- [Result] Kris MG, Camidge DR, Giaccone G, Hida T, Li BT, O'Connell J, Taylor I, Zhang H, Arcila ME, Goldberg Z, Janne PA. Targeting HER2 aberrations as actionable drivers in lung cancers: phase II trial of the pan-HER tyrosine kinase inhibitor dacomitinib in patients with HER2-mutant or amplified tumors. Ann Oncol. 2015 Jul;26(7):1421-7. doi: 10.1093/annonc/mdv186. Epub 2015 Apr 21. PMID 25899785
- [Result] Mazieres J, Peters S, Lepage B, Cortot AB, Barlesi F, Beau-Faller M, Besse B, Blons H, Mansuet-Lupo A, Urban T, Moro-Sibilot D, Dansin E, Chouaid C, Wislez M, Diebold J, Felip E, Rouquette I, Milia JD, Gautschi O. Lung cancer that harbors an HER2 mutation: epidemiologic characteristics and therapeutic perspectives. J Clin Oncol. 2013 Jun 1;31(16):1997-2003. doi: 10.1200/JCO.2012.45.6095. Epub 2013 Apr 22. PMID 23610105
- [Result] De Greve J, Teugels E, Geers C, Decoster L, Galdermans D, De Mey J, Everaert H, Umelo I, In't Veld P, Schallier D. Clinical activity of afatinib (BIBW 2992) in patients with lung adenocarcinoma with mutations in the kinase domain of HER2/neu. Lung Cancer. 2012 Apr;76(1):123-7. doi: 10.1016/j.lungcan.2012.01.008. Epub 2012 Feb 10. PMID 22325357
- [Result] Diaz R, Nguewa PA, Parrondo R, Perez-Stable C, Manrique I, Redrado M, Catena R, Collantes M, Penuelas I, Diaz-Gonzalez JA, Calvo A. Antitumor and antiangiogenic effect of the dual EGFR and HER-2 tyrosine kinase inhibitor lapatinib in a lung cancer model. BMC Cancer. 2010 May 11;10:188. doi: 10.1186/1471-2407-10-188. PMID 20459769
- [Result] Wang Y, Jiang T, Qin Z, Jiang J, Wang Q, Yang S, Rivard C, Gao G, Ng TL, Tu MM, Yu H, Ji H, Zhou C, Ren S, Zhang J, Bunn P, Doebele RC, Camidge DR, Hirsch FR. HER2 exon 20 insertions in non-small-cell lung cancer are sensitive to the irreversible pan-HER receptor tyrosine kinase inhibitor pyrotinib. Ann Oncol. 2019 Mar 1;30(3):447-455. doi: 10.1093/annonc/mdy542. PMID 30596880
- [Result] Zhou C, Li X, Wang Q, Gao G, Zhang Y, Chen J, Shu Y, Hu Y, Fan Y, Fang J, Chen G, Zhao J, He J, Wu F, Zou J, Zhu X, Lin X. Pyrotinib in HER2-Mutant Advanced Lung Adenocarcinoma After Platinum-Based Chemotherapy: A Multicenter, Open-Label, Single-Arm, Phase II Study. J Clin Oncol. 2020 Aug 20;38(24):2753-2761. doi: 10.1200/JCO.20.00297. Epub 2020 Jul 2. PMID 32614698